CLINICAL TRIAL: NCT07147127
Title: Anti-Citrullinated SR-A Peptide (Anti-csp)Antibody as a Biomarker for Rheumatoid Arthritis.
Brief Title: Anti-citrullinated SR-A Peptide (Anti-csp) Antibody as a Biomarker in Rheumatoid Arthritis (RA).
Status: Not yet recruiting | Type: Observational
Sponsor: Walaa sharif Eid Ahmed (Other)
Responsible Party: Sponsor-Investigator, Walaa sharif Eid Ahmed, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Anti-csp
Record Dates: First submitted 2025-08-09; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 27 seropositive patients according to results of rheumatoid factor and anticitrullinated antibodies.: 27 seronegative patients according to results of rheumatoid factor and anticitrullinated antibodies.
- 27 seronegative patients according to results of RF and ACCP

SUMMARY:
1. To measure serum level of anticitrullinated SR-A peptide antibody (anti-CSP) in RA patients compared to healthy controls .
2. To assess the diagnostic performance of anti-CSP for RA specifically seronegative RA patients.
3. To evaluate correlation of serum anti-CSP level with disease activity and functional disability scores in RA patients.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a common a chronic autoimmune disease that can lead to joint destruction, disability, and premature mortality .Early diagnosis is crucial for preventing long-term damage and disability.

Anticyclic citrullinated peptide antibody (anti-CCP) and rheumatoid factor (RF) are classical serological markers for the diagnosis of RA and have been integrated into the 2010 (ACR/EULAR) classification criteria for RA . However, they show a modest discriminating power. The sensitivity and specificity are 67% and 95% for antiCCP, and 69% and 85% for RF, respectively . Therefore, there is an unmet need to identify prospective diagnostic biomarkers for RA.

Several biomarkers have been identified in peripheral blood or synovial fluid of RA patients, including collagen, fibrinogen, vimentin, fibronectin, and α-enolase . Their posttranslational modification, in particular citrullination, is essential for the pathogenesis of RA. These citrullinated autoantigens could stimulate the secretion of autoantibodies, namely, anticitrullinated protein antibodies (ACPAs).

•Anti-CCP is one of the most common ACPAs. ACPAs demonstrate arthritogenic potential and perpetuate inflammation in RA through promoting innate immune cells binding ,complement system activation ,neutrophil extracellular traps (NETs) formation ,and osteoclasts activation . Moreover, accumulating experimental evidence revealed the contribution of the glycosylation changes of ACPAs to the systemic inflammation of RA .Several typical glycosylation patterns of ACPAs have also been identified in RA.

Macrophage scavenger receptor A (SR-A, CD204, MSR-1, SCARA1) is a kind of classical pattern recognition receptors (PRRs) primarily expressed on macrophages .Besides its role in innate immunity, accumulating evidence also indicated the functional significance of SR-A in adaptive immunity ,In a large-scale multicenter study, soluble SRA demonstrated a sensitivity of 66.41% and specificity of 91.45% for the diagnosis of RA, with positive predictive value (PPV) of 80.19% and negative predictive value (NPV) of 83.94%

. Detecting autoantibodies directed against CSP (anti- CSP) could therefore provide a new serological tool for RA diagnosis. These antibodies may not only enhance diagnostic accuracy particularly in patients who are seronegative for conventional markers but also shed light on novel mechanisms in RA pathophysiology

ELIGIBILITY:
Inclusion Criteria:

Adults (≥18 years old)

Exclusion Criteria:

Patients with other autoimmune or connective tissue diseases (e.g., SLE, SS) .

* Patients with chronic infections or malignancies .
* Patients less than18 years old .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seronegative and seropositive rheumatoid arthritis patients and health control group
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To assess the diagnostic performance of anti-Citrullinated SR-A peptide antibody (anti-csp) for rheumatoid arthritis specifically seronegative rheumatoid arthritis patients . | through study completion, an average of 1 year
To evaluate correlation of serum anti-CSP level with disease activity and functional disability scores in RA patients . | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xie Y, Wei C, Fu D, Zhang W, Du Y, Huang C, Liu S, Yao R, He Z, Zhang S, Jin X, Shen B, Cao L, Wang P, Fang X, Zheng X, Lin H, Wei X, Lin W, Bai M, Zhu D, Li Y, Ding Y, Zhu H, Ye H, He J, Su Y, Jia Y, Wu H, Wang Y, Xing D, Qiu X, Li Z, Hu F. Large-scale multicenter study reveals anticitrullinated SR-A peptide antibody as a biomarker and exacerbator for rheumatoid arthritis. Sci Adv. 2025 Jan 3;11(1):eadr8078. doi: 10.1126/sciadv.adr8078. Epub 2025 Jan 3. PMID 39752500